CLINICAL TRIAL: NCT00827255
Title: Physician's Evaluation of Cyclosporine Ophthalmic Emulsion 0.05%
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MA-RES-08-002
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Results first posted 2012-07-18 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients who received Restasis®: Patients who received Restasis® (cyclosporine ophthalmic emulsion 0.05%)
  Interventions: Drug: Cyclosporine Ophthalmic Emulsion 0.05%

INTERVENTIONS:
Drug: Cyclosporine Ophthalmic Emulsion 0.05% — One drop two times a day approximately 12 hours apart
  Other Names: RESTASIS®

SUMMARY:
The objective of this retrospective chart review is to evaluate the patient characteristics, treatment variations and efficacy of a second trial of Cyclosporine Ophthalmic Emulsion 0.05% therapy in chronic dry eye patients who were initially treated with Cyclosporine Ophthalmic Emulsion 0.05% but discontinued use after less than 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults >16 years of age
* Dry eye patients
* Subject with history of less than 12 weeks of initial RESTASIS® treatment
* Subject started second trial of RESTASIS® treatment prior to June 1, 2008
* First day of second trial of RESTASIS® started ≥ 4 weeks after the last day of previous RESTASIS® treatment

Exclusion Criteria:

* Patients with Contact Lens Intolerance
* Patients with Ocular Rosacea

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The medical charts of all chronic dry eye patients who discontinued their first trial of RESTASIS® after less than 12 weeks of treatment and who started a second trial of RESTASIS® prior to June 1, 2008 will be included in the review.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Mah F, Milner M, Yiu S, Donnenfeld E, Conway TM, Hollander DA. PERSIST: Physician's Evaluation of Restasis((R)) Satisfaction in Second Trial of topical cyclosporine ophthalmic emulsion 0.05% for dry eye: a retrospective review. Clin Ophthalmol. 2012;6:1971-6. doi: 10.2147/OPTH.S30261. Epub 2012 Nov 28. PMID 23226002

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Retrospective analysis. Patients may have been treated with Restasis® (cyclosporine ophthalmic emulsion 0.05%) in addition to other medications during the course of the study.
Period: Overall Study
Arm/Group | Patients Who Received Restasis®
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Who Received Restasis®
Number analyzed (Participants) | 35
Age, Customized [Number; unit: participants]
  <40 years | 7
  Between 40 and 49 years | 2
  Between 50 and 59 years | 8
  Between 60 and 69 years | 5
  Between 70 and 79 years | 11
  >=80 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Complete Clearing of Corneal Staining at Month 12
Description: Percentage of patients with complete clearing of corneal staining at month 12. Corneal staining is evaluated following administration of fluorescein dye into the eye. Complete clearing is defined as the absence of corneal staining.
Time Frame: Month 12
Population: ITT population, which consisted of all patients included in the study, with documented presence of corneal staining at baseline. For this outcome measure, a total of 18 patients had documented corneal staining at baseline.
Measure: Number; unit: Percentage of Patients
Arm/Group | Patients Who Received Restasis®
Number analyzed (Participants) | 18
Percentage of Patients | 33.3

2. Secondary Outcome: Schirmer's Test at Month 12
Description: Schirmer's test at month 12. The Schirmer's tear test is performed on the eye with or without anesthesia (numbing eye drop). The amount of tears produced by the eye in 5 minutes is measured in millimeters by means of a graduated paper scale. Data not reported due to limited number of patients with Schirmer's test data recorded.
Time Frame: Month 12
Population: ITT population, which consisted of all patients included in the study with Schirmer's testing data available at baseline. Data not reported due to limited number of patients with Schirmer's test data recorded.
Arm/Group | Patients Who Received Restasis®
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Serious adverse events and adverse events were not collected directly as this was a retrospective study.
Arm/Group | Patients Who Received Restasis®
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo